CLINICAL TRIAL: NCT03945331
Title: Characterization of Transcutaneous and Epidural Spinal Stimulation for Enabling Motor Function in Humans With Motor Complete Paraplegia
Brief Title: Transcutaneous and Epidural Spinal Stimulation for Enabling Motor Function in Humans With Motor Complete Paraplegia
Acronym: TransEpi
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 disrupted interventions irrecoverably.
Sponsor: Mayo Clinic (Other)
Collaborators: Minnesota Office of Higher Education (Other Government)
Responsible Party: Principal Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18-011086
Record Dates: First submitted 2019-04-28; First posted 2019-05-10 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Paraplegia, Spinal; Paraplegia, Complete; Paraplegia; Traumatic
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- TESS (Experimental): Transcutaneous Electrical Spinal Stimulation (TESS), used during all training sessions.
  Interventions: Device: Transcutaneous spinal cord stimulator
- EES (Experimental): TESS, used during the initial 6-month training period, followed by Epidural Electrical Stimulation (EES) during the final 6-month training period.
  Interventions: Device: Transcutaneous spinal cord stimulator; Device: Epidural spinal cord stimulation system

INTERVENTIONS:
Device: Transcutaneous spinal cord stimulator — DS8R Electrical Stimulator For Human Research
Device: Epidural spinal cord stimulation system — Spectra WaveWriter Epidural Spinal Cord Stimulator System with CoverEdge 32 Electrode Surgical Lead
  Arms: EES

SUMMARY:
The purpose of this study is to compare transcutaneous electrical spinal stimulation (TESS) and epidural electrical stimulation (EES); in particular, the motor activity enabled by each method and the potential health benefits of each method.

ELIGIBILITY:
Inclusion Criteria

* Spinal cord injury due to trauma located between the seventh cervical and tenth thoracic vertebrae
* American Spinal Injury Association grading scale of A or B (at least 4 each of A and B) below the level of SCI
* Intact spinal reflexes below the level of SCI
* At least 1-year post-SCI
* At least 22 years of age
* Willing to use medically acceptable methods of contraception, if female and of child-bearing potential

Exclusion Criteria

* Currently a prison inmate, or awaiting trial, related to criminal activity
* Pregnancy at the time of enrollment
* DEXA t score <-3.5 at spine and femur head
* History of chronic and/or treatment resistant urinary tract infection
* Unhealed decubitus ulcer
* Unhealed skeletal fracture
* Untreated clinical diagnosis of depression
* Presence of joint contractures or an Ashworth spasticity score of 4
* Active anti-spasticity medication regimen within 3 months prior to study enrollment
* Presence of transcranial magnetic stimulation-evoked potentials in leg muscles
* Non MRI-compatible implanted medical devices.
* Undergoing, or planning to undergo, diathermy treatment
* Active participation in another interventional clinical trial
* Presence of conditions or disorders which require MRI monitoring
* For EES cohort subjects, a history of coagulopathy or other significant cardiac or medical risk factors for surgery
* Current use of a ventilator
* Clinically diagnosed cardiopulmonary complications such as chronic obstructive pulmonary disease, cardiac failure, or heart arrhythmia that contraindicate changes in body position such as supine-to-sit-to-stand activities, prolonged standing, or stepping
* Mass > 113 kg (250 pounds)
* History of frequent hypotension characterized by light headedness, or loss of consciousness
* History of frequent hypertension characterized by headache, or bradycardia
* History of frequent, severe, autonomic dysreflexia
* Any illness or condition which, based on the research team's assessment, will compromise with the patient's ability to comply with the protocol, patient safety, or the validity of the data collected during this study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Kinematics | Baseline, Month 3, Month 6, End of Month 7, Month 10, Month 13
  Change in measurements of joint angles using video-based, inertial measurement, and/or electromagnetic markers.
Electromyography | Baseline, Month 3, Month 6, End of Month 7, Month 10, Month 13
  Change in measurements of electrical activity at major muscle groups below the level of injury.
Foot pressure | Baseline, Month 3, Month 6, End of Month 7, Month 10, Month 13
  Change in measurements of foot pressure through shoe-insole pressure sensors.
Somatosensory evoked potentials | Baseline, Month 6, End of Month 7, Month 13
  Change in measurements of change in conduction in the peripheral nerves, cervical and lumbosacral spinal cord, deep brain structures, and sensory cortex, through surface electrodes.
Transcranial magnetic stimulation motor evoked potentials | Baseline, Month 6, End of Month 7, Month 13
  Change in measurements of stimulus intensity required to elicit muscle responses in muscle groups known to elicit optimal motor evoked potential responses, both above and below the level of injury.
Monosynaptic spinal reflex testing | Baseline, Month 6, End of Month 7, Month 13
  Change in measurements of stimulation intensity H and F wave thresholds and maximal responses through surface electrodes.
Trunk stability | Baseline, Month 3, Month 6, End of Month 7, Month 10, Month 13
  Change in measurements of trunk stability using the modified functional reach test (mFRT).
Injury severity: American Spinal Injury Association Impairment Scale (AIS) | Baseline, Month 6, End of Month 7, Month 13
  Change in measurements of impairment of sensory and motor functions using the American Spinal Injury Association Impairment Scale (AIS). Individuals are classified from A" (complete spinal cord injury) to "E" (normal function). 28 dermatomes and 10 key muscles are assessed bilaterally. Results are summed to produce overall sensory and motor scores and are used in combination with evaluation of anal sensory and motor function as a basis for the determination of AIS classification. Sensory scores are rated 0 (sensation absent) to 2 (normal), bilaterally for each of 28 dermatomes. Muscle function is rated 0 (total paralysis) to 5 (active movement, full range of motion against significant resistance) for each myotome. Upper Extremity Motor Subscores and Lower Extremity Motor Subscores are each scored from 0 to 50; the ASIA Motor Score is scored from 0 to 100. The presence of anal sensation and voluntary anal contraction are assessed as a yes/no.

SECONDARY OUTCOMES:
Bowel function | Baseline, Month 6, Month 13
  Change in measurements of bowel function utilizing anorectal manometry.
Bladder function | Baseline, Month 6, Month 13
  Change in measurements of bladder function utilizing a urodynamic test consisting of a filling phase and a voiding phase cystometrogram along with perineal patch muscle electromyography.
Spasticity | Baseline, Month 3, Month 6, End of Month 7, Month 10, Month 13
  Change in measurements of spasticity using the Modified Ashworth Scale (MAS), an assessment which measures resistance during passive soft-tissue stretching of bilateral hip flexors, extensors, adductors, and abductors, knee extensors and flexors, and ankle plantarflexors and dorsiflexors. Scoring is scaled from 0 (no increase in muscle tone) to 4 (affected part[s] rigid in flexion or extension), with higher scores indicating more spasticity.
Bone mineral density | Baseline, Month 6, Month 13
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in bone mineral content and bone density.
Body composition - body fat mass | Baseline, Month 6, End of Month 7, Month 13
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in regional and total body fat mass.
Body composition - lean mass | Baseline, Month 6, End of Month 7, Month 13
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in regional and total lean mass.
Body composition - android and gynoid fat percentage | Baseline, Month 6, End of Month 7, Month 13
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in regional and total android and gynoid fat percentage.
Body composition - android and gynoid fat ratio | Baseline, Month 6, End of Month 7, Month 13
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in regional and total android to gynoid fat ratio.
Body composition - bone mass | Baseline, Month 6, End of Month 7, Month 13
  Measurement by dual-energy x-ray absorptiometry (DXA) of change in regional and total bone mass.
Knee cartilage health | Baseline, Month 6; Month 13 for TESS cohort only
  Assessment of change in knee cartilage breakdown using the modified Outerbridge classification or the International Cartilage Repair Society classification, utilizing magnetic resonance imaging (MRI).
Metabolics - CBC | Baseline, Month 6, End of Month 7, Month 13
  Measurement of changes in complete blood count with differential.
Metabolics - glucose | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in fasting glucose value.
Metabolics - total cholesterol | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in total cholesterol value.
Metabolics - HDL cholesterol | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in HDL cholesterol value.
Metabolics - calculated LDL cholesterol | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in calculated LDL cholesterol value.
Metabolics - triglycerides | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in triglycerides value.
Metabolics - non-HDL cholesterol | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in non-HDL cholesterol value.
Spinal structural integrity | Baseline
  Assessment of structural integrity via computerized tomography (CT).
Injury severity and potential for spared tissue | Baseline
  Evaluation of severity and possibility of discomplete injury despite complete loss of motor function via MRI.
Stimulator array location and migration (EES cohort only) | End of Month 7, Month 13
  Evaluation of current array location via CT.
Patient-reported bowel function (1) | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in bowel function using the Neurogenic Bowel Dysfunction Score. Answers to qualitative questions are rated from 0 to 5, with a higher number indicating more problematic symptoms, and totaled for a score which categorizes severity of neurogenic bowel symptoms.
Patient-reported bowel function (2) | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in bowel function using the International Spinal Cord Injury Bowel Function Basic Data Set (v2.0). Answers to qualitative questions are rated from 0 to 13, with a higher number indicating more problematic symptoms, and totaled for a score which categorizes neurogenic bowel dysfunction.
Patient-reported bladder function (1) | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in bladder function using the Neurogenic Bladder Symptom Score. Answers to qualitative questions are rated from 0 to 5, with a higher number indicating more problematic symptoms, and totaled for a score which categorizes severity of neurogenic bladder symptoms.
Patient-reported bladder function (2) | Baseline, Month 6, End of Month 7, Month 13
  Assessment of change in bowel function using the International Spinal Cord Injury Urodynamic Basic Data Set. Data from various urodynamic variables are aggregated into a single-page format for an abstract overview of bladder dysfunction.
Male patient-reported sexual function (1) | Baseline, Month 6, End of Month 7, Month 13
  Assessment of change in sexual function using the International Spinal Cord Injury Male Sexual Function Basic Data Set (v2.0). Data from various male sexual function variables are aggregated into a single-page format for an abstract overview of male sexual dysfunction.
Male patient-reported sexual function (2) | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in erectile dysfunction using the Sexual Health Inventory for Men (SHIM). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better erectile function, and totaled for a score which categorizes severity of erectile dysfunction.
Male patient-reported sexual function (3) | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in erectile dysfunction using the International Index for Erectile Function (IIEF). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better erectile function, and totaled for a score which categorizes severity of erectile dysfunction.
Female patient-reported sexual function (1) | Baseline, Month 6, End of Month 7, Month 13
  Assessment of change in sexual function using the International Spinal Cord Injury Female Sexual and Reproductive Function Basic Data Set (v2.0). Data from various female sexual and reproductive function variables are aggregated into a single-page format for an abstract overview of female sexual and reproductive dysfunction.
Female patient-reported sexual function (2) | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change in sexual function using the Female Sexual Function Index (FSFI). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better sexual function, and totaled for a score which categorizes severity of sexual dysfunction.
Patient-reported quality of life (1): Spinal Cord Injury Secondary Conditions Scale (SCI-SCS) | Baseline, Month 6, End of Month 7, Month 13
  Measurements of change to quality of life as measured by the Spinal Cord Injury Secondary Conditions Scale (SCI-SCS). Answers to qualitative questions regarding patient activities, independence, and overall quality of life are rated from 0 to 3, with a higher number indicating more significant or chronic problems, and totaled for a score which categorizes patient quality of life.
Patient-reported quality of life (2): World Health Organization Quality of Life Questionnaire (WHOQOL-BREF) | Baseline, Month 6, End of Month 7, Month 13
  Measurement of change to quality of life as measured by the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF). Answers to qualitative questions regarding patient activities, independence, and overall quality of life are rated from 1 to 5, with a higher number indicating a higher concurrence or frequency related to the item in question, and totaled for a score which categorizes patient quality of life.

OTHER OUTCOMES:
Volitional movement (1) | 1 year
  Measurement of change in volitional movement through recordings of training time in minutes.
Volitional movement (2) | 1 year
  Measurement of change in volitional movement through recordings body weight support measured as a percentage of total body weight supported.
Volitional movement (3) | 1 year
  Measurement of change in volitional movement through recordings of speed in miles per hour.
Volitional movement (4) | 1 year
  Measurement of changes in volitional movement through recordings of assistive devices used.
Volitional movement (5) | 1 year, for TESS cohort only
  Measurement of changes in volitional movement through recordings of stimulator electrode location.
Volitional movement (6) | 1 year
  Measurement of changes in volitional movement through recordings of stimulator intensity, measured in milliamps per volt.
Volitional movement (7) | 1 year
  Measurements of changes in volitional movement through recordings of stimulator frequency measured in Hertz.
Volitional movement (8) | 1 year
  Measurement of changes in volitional movement through recordings of pulse width, measured in microseconds.
Overground ambulation [as appropriate to the subject] (1) | 1 year
  Measurement of changes in overground mobility as measured by the SCI Functional Ambulation Inventory. Trainer ratings of various gait parameters and criteria are rated from 0 to 5, with a higher number indicating better walking mobility, and totaled for a score which characterizes overall functional ambulation.
Overground ambulation [as appropriate to the subject] (2) | 1 year
  Measurement of changes in overground mobility as measured by the Modified 6 Minute Walk Test. Trainers will assess the distance in meters which the subject can cover in 6 minutes, with a greater distance characterizing better overground mobility.
Overground ambulation [as appropriate to the subject] (3) | 1 year
  Measurement of changes in overground mobility as measured by the Modified Timed Up and Go test. Trainers will assess the time it takes, in minutes and seconds, for the subject to stand from a chair, move out to a 3 meter distance, return to the chair and sit down. Less time will characterize better overground mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin D. Zhao, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials